CLINICAL TRIAL: NCT06860074
Title: The Effect of Sustainable Environmental Health Program Planned for High School Students on Environmental Sensitivity, Sustainable Environmental Awareness, Environmental Attitudes and Behaviors: a Randomized Controlled Trial
Brief Title: Sustainable Environmental Health Program for Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Feyza Bardak, Principal Investigator, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E- 87432956-050.99-755267
Record Dates: First submitted 2025-02-14; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Health Behavior; Sustainability; Environment
Keywords: Environment; Environmental Health; Adolescent
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Masking will not be possible due to the method of application of this study. However, the data collector, statistician and reporting will be masked during the research process. In the research process, pre-test data will be collected by the teachers working in the study school. The post-test data will be collected by another researcher (a researcher trained in the data collection form and trained in the field of nursing).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): No Intervention
- Intervention Group (Experimental): Sustainable Environmental Health Programs
  Interventions: Behavioral: Sustainable Environmental Health Programs

INTERVENTIONS:
Behavioral: Sustainable Environmental Health Programs — * Sustainable Future: Environment, Ecological Balance and Health,
  * Ecological Balance and Pollution: Protecting Environmental Health
  * Ecological Balance and Environmental Health
  * A New Life for Waste: A Sustainable Future with Recycling
  * Environmental Behaviors
  * Recycling for Street Animals: A Shed Construction Project
  Arms: Intervention Group

SUMMARY:
The research will be conducted to determine the effect of the sustainable environmental health program on environmental sensitivity, sustainable environmental awareness, environmental attitudes and behaviors in high school students. The purpose of this study is to develop and sustain environmental sensitivity, sustainable environmental awareness, environmental attitudes and behaviors in high school students with the Sustainable Environmental Health Program.

DETAILED DESCRIPTION:
Environmental health has direct and indirect impacts on ecosystem balance and human health. Among the consequences of adverse environmental conditions, non-communicable diseases, including ischaemic heart disease, chronic respiratory diseases and cancers, are the most common. Situations such as environmental pollution, climate change, deforestation and loss of biodiversity that negatively affect environmental health are important public health problems. Protection and improvement of environmental health is very important in terms of sustainable development goals.

Many institutions and organisations carry out studies within the scope of sustainable development goals. The basis of the studies carried out in this context is to improve environmental behaviours. The studies carried out in the field of health include public health studies to protect and improve environmental health. In addition, environmental sensitivity, sustainable environmental awareness and environmental attitude are very important in the development and sustainability of environmental behaviours. The development of environmental sensitivity, awareness, attitudes and behaviours in adolescence is important for individual, social and environmental health now and in the future.

Intervention activities carried out to develop environmental awareness, consciousness, attitude and behaviours are interactive interventions such as message content, interaction with nature, education through presentation, cinevision, peer education and puzzle activities.

It is seen that there are cognitive, affective and behavioural changes within the scope of intervention activities. However, when the selected intervention is based on a single teaching method, its effectiveness differs due to the difference in individual perception levels. Combining different intervention activities can eliminate the differences in individual perception levels. The programme prepared by considering different intervention techniques in adolescence is important to develop environmental sensitivity, sustainable environmental awareness and environmental attitude and to ensure the formation of environmental behaviours. For this reason, this study examines the effect of the sustainable environmental health programme on the development of environmental sensitivity, sustainable environmental awareness, environmental attitudes and behaviours in high school students.

ELIGIBILITY:
Inclusion Criteria:

1. Studying in the 9th grade,
2. Being able to speak and understand Turkish,
3. Parental consent for participation,
4. Volunteering to participate in the research

Exclusion Criteria:

1. Having received previous education on environmental health,
2. Transported education
3. Boarding education and training

Ages: 13 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 98 (Estimated)
Dates: Start 2025-03-02 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Environmental Behavior | 3 months
  Environmental Behavior Scale was originally developed by Ardahan (2022). The scale consists of three sub-dimensions as "Sharing in the Family", "Behavior at Home" and "Sharing at School", and a total of 13 items. The scale is evaluated on a five-point Likert scale, rated as "Strongly agree", "Agree", "Undecided", "Disagree" and "Strongly disagree". The internal validity and variance of the scale; Cronbach's Alpha coefficient was stated as 0.888 and the variance explained by the scale was 66.85%. It was stated that the smallest value that can be taken from the scale is 13 and the largest value is 65.

SECONDARY OUTCOMES:
Attitude Scale Towards Environmental Problems | 3 months
  The scale developed has a total of 22 items and a four-factor structure. The scale is rated in a five-point Likert type. The factors in the scale are; Negative Affective Component, Cognitive Component, Behavioral Component and Positive Affective Component, respectively. The total Cronbach alpha value of the scale is .88 and the Cronbach alpha values of the factors are .84, .78, .73 and .70, respectively.
Sustainable environmental awareness | 3 months
  The Sustainable Environmental Awareness Scale was prepared by utilizing the course contents in the education-training curriculum, aiming to reach the information about what students do under certain conditions. The scale is single-dimensional, has a total of 10 items and a 3-point Likert level. In each item in the scale, the desired situation is calculated as three points, the partially desired situation as two points and the undesirable situation as one point. The highest score that can be obtained from the scale is 30 (3x10), the lowest score is 10 (1x10), and the average score of the scale is 20. When the factor loadings of the scale are examined, it is stated that they vary between 0.585 and 0.735 and the total Cronbach alpha value is 0.87. In addition, the scale explains 45.87% of the total variance
Environmental Sensitivity | 3 months
  The Environmental Awareness Questionnaire consists of 24 questions. In the questionnaire, the scale items were prepared with a three-degree answer feature consisting of "Always", "Sometimes" and "Never" options in order to determine the sensitivity towards air pollution, water pollution, soil pollution, green area problems and population growth and ecological balance. The alpha reliability coefficient of the questionnaire was found to be 0.81 in the original study (α). Factor analysis test was used for the structural validity of the sub-factors and as a result of the factor analysis conducted, it was determined by the developers that all 24 items determined for the trial form were suitable. Evaluation was made by giving a total score between the lowest 24 and the highest 72 points, with those who answered "always" receiving 3 points, those who answered "sometimes" receiving 2 points, and those who answered "never"

IPD SHARING:
Plan to Share IPD: Undecided